CLINICAL TRIAL: NCT05597488
Title: EUS Guided Portal-systemic Pressure Gradient Measurement to Predict Treatment Response and Outcomes of Varices to Endoscopic Variceal Ligation in Patients With Chronic Hepatitis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Anthony Teoh, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022.088
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Cirrhosis Portal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EUS guided portal pressure gradient measurement (Experimental): At index OGD, the presence and severity of OV, GV and portal hypertensive gastropathy would be recorded. After endoscopic treatment of varices, recruited patients would undergo 1st measurement of EUS-PPG within 10-14 days after index OGD. The patients would then be enrolled into a variceal surveillance program and be started on B-blockers if not already prescribed. The patients would then be scheduled for another follow-up OGD at 3 months with measurement of the 2nd EUS-PPG. Finally, a third follow-up OGD and EUS-PPG would be performed in 1-year after 1st EUS-PPG. Endoscopic findings attributed to chronic cirrhosis would be assessed in the 3 months and 1 year OGD and the presence and severity of OV, GV and portal hypertensive gastropathy would be recorded.
  Interventions: Device: EUS guided portal pressure gradient measurement

INTERVENTIONS:
Device: EUS guided portal pressure gradient measurement — EUS-guided PPGM is performed under monitored anaesthesia. The linear array echoendoscope is passed from the mouth into the stomach and duodenum, as with a standard exam. Under endoscopic ultrasound guidance, a 25 gauge EUS needle (Echotip, Cook Medical, USA) primed with heparin 100 USP/ml is then placed across the stomach or duodenal wall and through the liver parenchyma into the portal vein (Figure 3). A pressure measurement is then obtained from the compact pressure transducer attached to the handle of the needle (Figure 4). Three separate measurements are made with re-priming of heparin (less than 0.5 ml). The needle is then removed from the portal vein and liver, if necessary. The process is repeated for the hepatic vein (Figure 5). The EUS - PPG is calculated by subtracting the average of the three hepatic vein pressure measurements from the average of the 3 direct portal vein pressure measurements.

SUMMARY:
The aim of the current study is to assess if EUS-PPGM could predict the treatment response and outcomes of varices to endoscopic variceal ligation (EVL) in patients with chronic hepatitis. The hypothesis is that a high EUS-PPGM value at 3 months correlates with the presence of varices requiring EVL in patients that have received primary or secondary variceal prophylaxis on 1 year follow-up upper endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 75 years old
* Informed consent available
* Suffering from chronic hepatitis induced cirrhosis
* Suffering from oesophageal varices and received EVL as a result of

  1. Primary variceal prophylaxis during a variceal surveillance program on oesophagogastroduodenoscopy (OGD) or
  2. Secondary variceal prophylaxis after EVL in patients with active oesophageal variceal bleeding
* Or bleeding gastric varices that have received endoscopic canoacrylate injection

Exclusion Criteria:

* Medical Child-Pugh Class C Uncorrected platelet count <50,000 INR > 1.5 (natural) History of hepatic encephalopathy Current or history of hepatocellular carcinoma
* Anatomical Main portal vein thrombosis Anatomic alterations of the hepatic vasculature that prevent access to the portal vein or intrahepatic portion of the hepatic veins (identified at screening and/or during the endoscopic procedure).

Previous history of spontaneous bacterial peritonitis within the previous three months Portopulmonary hypertension Cardiac decompensation

- Endoscopically Confirmed Exclusion Criteria Presence of ascites in the path of the needle that prevents apposition of the gastrointestinal tract and liver.

Presence of gastric or duodenal ulcers, dieulafoy's lesion or cancers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Presence or absence of varices requiring EVL on 1 year follow-up upper endoscopy | 1 year
  The number of patients with a high EUS-PPGM at 3 months will be correlated with the presence or absence of varices requiring EVL on 1 year follow-up upper endoscopy.

SECONDARY OUTCOMES:
Other outcome measurements | 1 year
  The value of Day 0, 3 months or 1year EUS-PPG would be correlated with the severity of cirrhosis, re-bleeding, number of sessions of repeated EVL and mortality at 1 year. Safety of the procedure would also be assessed as 30-day adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No